CLINICAL TRIAL: NCT06805617
Title: A Phase 2 Trial of Ivonescimab for Patients With Advanced, Metastatic Salivary Gland Cancers (I-MAC)
Brief Title: A Phase 2 Trial of Ivonescimab for Patients With Advanced, Metastatic Salivary Gland Cancers
Acronym: I-MAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Glenn J. Hanna (Other)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Glenn J. Hanna, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-746
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Salivary Gland Cancer; Advanced Salivary Gland Carcinoma; Metastatic Salivary Gland Cancer; Adenoid Cystic Carcinoma
Keywords: Salivary Gland Cancer; Salivary Gland Carcinoma; Metastatic Salivary Gland Cancer; Adenoid Cystic Carcinoma
MeSH Terms: conditions — Salivary Gland Neoplasms; Carcinoma, Adenoid Cystic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Adenoid Cystic Carcinoma (Experimental): Approximately 11 participants will be enrolled to this cohort in the first stage of recruitment. If there are ≤2 participants (out of 22) with responses to the therapy, the accrual to the study will be stopped. If there are >2 participants with response, accrual will continue. Enrolled participants will complete:
  * Baseline visit
  * Imaging tests every 9 weeks
  * Cycle 1 through End of Treatment (21 day cycles)
    --Day 1: Predetermined dose of Ivonescimab 1x daily.
  * End of treatment visit with imaging
  * Follow up: every 12 weeks
  Interventions: Drug: Ivonescimab
- Cohort 2: Non-Adenoid Cystic Carcinoma Salivary Gland Carcinoma (Experimental): Approximately 11 participants will be enrolled to this cohort in the first stage of recruitment. If there are ≤2 participants (out of 22) with responses to the therapy, the accrual to the study will be stopped. If there are >2 participants with response, accrual will continue. Enrolled participants will complete:
  * Baseline visit
  * Imaging tests every 9 weeks
  * Cycle 1 through End of Treatment (21 day cycles)
    --Day 1: Predetermined dose of Ivonescimab 1x daily.
  * End of treatment visit with imaging
  * Follow up: every 12 weeks
  Interventions: Drug: Ivonescimab

INTERVENTIONS:
Drug: Ivonescimab — An immunoglobulin (Ig) G1 monoclonal antibody (mAb), single-use vial, via intravenous (into the vein) infusion per protocol.
  Other Names: SMT112; AK112

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of Ivonescimab in participants with advanced, metastatic salivary gland cancers.

The name of the study drug involved in this study is:

-Ivonescimab (a type of antibody)

DETAILED DESCRIPTION:
This is phase 2, open-label, non-randomized study is to investigate Ivonescimab in participants with incurable, recurrent or metastatic salivary gland carcinomas (SGC). Ivonescimab is expected to treat salivary gland cancer by blocking or slowing cancer cell growth

The U.S. Food and Drug Administration (FDA) has not approved Ivonescimab as a treatment for advanced, metastatic salivary gland cancer but it has been used as treatment for lung cancer.

The study procedures include screening for eligibility, in-clinic visits, X-rays, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, or Positron Emission (PET) scans Computerized, blood tests, urine tests, and tumor biopsies.

Participants will be in this study for approximately 3 years including follow-up after active study treatment.

It is expected that about 35 people will take part in this research study.

Summit Therapeutics, a pharmaceutical company, is supporting this research study by providing funding for the research and the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed salivary gland carcinoma (any histologic subtype, including ACC) with evidence of recurrent, metastatic, or advanced, unresectable disease.
* Willing to provide tumor tissue from a diagnostic biopsy or prior surgery if deemed safe and feasible by the investigator.
* Age 18 years or older at the time of consent. There is no upper age limit restriction in an effort to include patients across the lifespan.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Participant must have organ and marrow function as defined below within 14 days prior to study registration:

  * Absolute neutrophil count (ANC) ≥1000/mcL
  * Hemoglobin ≥8.5 g/dL (with no blood transfusions within 7 days of start of therapy)
  * Platelets ≥100,000/mcL
  * Liver function:

    * Serum total bilirubin (T-bili) ≤1.5× upper limit of normal (ULN); for patients with liver metastases or confirmed/suspected Gilbert syndrome, T-bili ≤3× ULN
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5× ULN; for patients with liver metastases, AST and ALT ≤5× ULN
  * Creatinine Within normal limits, or Creatinine clearance (CrCl) ≥50 mL/min using the Cockcroft-Gault formula or estimated glomerular filtration rate (eGFR) value ≥50 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (adjustment by BSA is not required for eGFR)
  * Urine protein: Urine protein <2+ or 24-hour urine protein quantification <1.0 g
  * Coagulation:prothrombin time (PT) or international normalized ratio (INR) ≤1.5× ULN, and partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) ≤1.5× ULN (unless abnormalities are unrelated to coagulopathy or coagulation)
* Participants must have documentation of a new or progressive lesion on a radiologic imaging study performed within 12 months prior to study registration (progression of disease over any interval is allowed) and/or new or worsening disease-related symptoms within 12 months prior to study registration. This assessment is performed by the treating investigator. Evidence of progression by RECIST v1.1 criteria is not required.
* Participants must have at least one RECIST v1.1 measurable non-CNS based lesion, as defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) ≥1 cm with CT scans or MR imaging.
* Prior systemic therapy: At least 2 weeks must have elapsed since the end of prior chemotherapy, biological agents (3 weeks for anti-cancer monoclonal antibody containing regimens) or any investigational drug product, with adequate recovery of treatment-related toxicity to NCI CTCAE Version 5.0 grade ≤1 (or tolerable grade 2) or back to baseline (except for alopecia or neuropathy). Any number of prior therapies for recurrent/metastatic SGC are permitted except receipt of a prior oral VEGFR TKI or anti-PD-1 therapy; but prior therapy for recurrent/metastatic SGC is not required for participation.
* Ability to understand and the willingness to sign a written informed consent document.
* Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 14 days of study registration. Female subjects of childbearing potential should have a negative urine or serum pregnancy test repeated within 72 hours prior to receiving the first dose of study medication.
* Female patient of childbearing potential having sex with an unsterilized male partner must agree to use a highly effective method of contraception from the beginning of screening until 120 days after the last dose of the Ivonescimab.
* Unsterilized male patient having sex with a female partner of childbearing potential must agree to use an effective method of contraception from the beginning of screening until Day 120 after the last dose of Ivonescimab.

Exclusion Criteria:

* Participant has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment) and have no evidence of new or enlarging brain metastases.
* Concurrent administration of other cancer specific therapy or investigational agents during the course of this study is not allowed.
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant or lactating women as the effects of the investigational therapy (ivonescimab) on the developing human fetus are unknown.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer, and low- risk prostate adenocarcinoma being managed with active surveillance. A history of another separate malignancy in remission without evidence of active disease in the last 2 years is permitted.
* Existing significant autoimmune conditions. Patients with a history of Hashimoto thyroiditis who are stable on replacement hormone therapy are not excluded. Patients cannot be on long-term (>4 weeks) corticosteroids at doses exceeding prednisone 10 mg daily (or its equivalent).
* Major surgical procedures or serious trauma within 4 weeks prior to starting therapy or plans for major surgical procedures within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) are permitted.
* History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to the start of therapy, including but not limited to:

  * a. Gastrointestinal bleeding
  * b. Hemoptysis (defined as coughing up ≥0.5 teaspoon of fresh blood or small blood clots). Note: transient hemoptysis associated with diagnostic bronchoscopy is allowed.
  * c. Significant nasal bleeding/epistaxis (bloody nasal discharge is allowed)
  * d. Need for therapeutic anticoagulant therapy within 14 days prior to the start of therapy.
* Current hypertension with systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg after oral antihypertensive therapy.
* History of major diseases , specifically:

  * a. Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] classification ≥ grade 2) or vascular disease (eg, aortic aneurysm at risk of rupture) that required hospitalization within 12 months prior to randomization, or other cardiac impairment that may affect the safety evaluation of the study drug (eg, poorly controlled arrhythmias, myocardial ischemia)
  * b. History of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months before randomization
  * c. History of arterial thromboembolic event, venous thromboembolic event of Grade 3 and above as specified in National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 6 months prior to randomization
  * d. Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks before randomization
  * e. History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to randomization
* Imaging during the screening period shows that the patient has:

  * a. Radiologically documented evidence of major blood vessel invasion or encasement by cancer (per the judgment of the treatment investigator)
  * b. Radiographic evidence of intratumor cavitation (per the judgment of the treating investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  ORR was defined as the percentage of participants achieving complete response (CR) and partial response (PR) on treatment based on RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Median Progression-Free Survival (PFS) | Up to 2 years
  Progression-Free Survival (PFS) based on Kaplan-Meier method is defined as the time from registration to the earlier of first progression, or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
Median Overall Survival (OS) | Up to 5 years
  Overall Survival (OS) based on Kaplan-Meier method is defined as the time from registration to death due to any cause or censored at date last known alive.
Duration of Response (DOR) | Up to 2 years
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause. Participants without events reported are censored at the last disease evaluation).
Duration of Response [Cohort 1] | Up to 2 years
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause. Participants without events reported are censored at the last disease evaluation).
Duration of Response [Cohort 2] | Up to 2 years
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause. Participants without events reported are censored at the last disease evaluation).
To evaluate safety and toxicity (CTCAE v5.0) | Up to 2 years
  Adverse events will be collected from the time of the first dose of study treatment, through the study and within 90 days of the last study intervention. Adverse events will be classified and graded according to the CTCAE v.5.0. Frequencies and/or rates of adverse events will be summarized among patients who begin protocol therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu